CLINICAL TRIAL: NCT02118649
Title: Enhancing Behavior and Brain Response to Visual Targets Using a Computer Game
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-10788
Record Dates: First submitted 2014-04-05; First posted 2014-04-21 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Game (Experimental): Participants will play a video game directing their gaze to on-screen targets.
  Interventions: Behavioral: Game

INTERVENTIONS:
Behavioral: Game

SUMMARY:
Participants will play a computer game that is controlled by their gaze patterns and designed to direct attention their attention to specific on-screen targets. Visual attention to targets will be rewarded. Both visual behavior and brain response will be recorded during game play.

It is hypothesized that that, over the course of the game, relative to baseline, participants will show (a) increased looking to targets, (b) decreased response time to targets, and (c) enhanced, more efficient neural response to visual cues. It is hypothesized that clinical variability will associate with visual attention and brain response.

ELIGIBILITY:
Inclusion Criteria:

* Able to participate in an eye-tracking experiment
* Able to participate in an EEG experiment

Exclusion Criteria:

* Sensory or physical impairment that would preclude completion of protocol
* Participants taking prescription medications that may affect cognitive processes
* Participants reporting significant head trauma or history of seizures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
EEG brain response to targets | Measures will be recorded for the duration of their visit, an expected average of 3 hours.

SECONDARY OUTCOMES:
Visual attention to targets as measured by eye-tracking | Measures will be recorded for the duration of their visit, an expected average of 3 hours.
Social Responsiveness Scale, Second Edition | Measures will be collected during visit, an expected average of 3 hours.
Autism Diagnostic Observation Schedule | Measures will be collected during visit, an expected average of 3 hours.
Differential Abilities Scale | Measures will be collected during visit, an expected average of 3 hours.
Vineland Adaptive Behavior Scales, Second Edition | Measures will be collected during visit, an expected average of 3 hours.
Social Anxiety Scale for Children, Revised | Measures will be collected during visit, an expected average of 3 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Hutt C, Ounsted C. The biological significance of gaze aversion with particular reference to the syndrome of infantile autism. Behav Sci. 1966 Sep;11(5):346-56. doi: 10.1002/bs.3830110504. No abstract available. PMID 5970485
- [Background] Senju A, Tojo Y, Yaguchi K, Hasegawa T. Deviant gaze processing in children with autism: an ERP study. Neuropsychologia. 2005;43(9):1297-306. doi: 10.1016/j.neuropsychologia.2004.12.002. Epub 2005 Jan 24. PMID 15949514
- [Background] Senju A, Yaguchi K, Tojo Y, Hasegawa T. Eye contact does not facilitate detection in children with autism. Cognition. 2003 Aug;89(1):B43-51. doi: 10.1016/s0010-0277(03)00081-7. PMID 12893128
- [Background] Tanaka JW, Wolf JM, Klaiman C, Koenig K, Cockburn J, Herlihy L, Brown C, Stahl S, Kaiser MD, Schultz RT. Using computerized games to teach face recognition skills to children with autism spectrum disorder: the Let's Face It! program. J Child Psychol Psychiatry. 2010 Aug;51(8):944-52. doi: 10.1111/j.1469-7610.2010.02258.x. PMID 20646129
- [Background] Tanaka JW, Wolf JM, Klaiman C, Koenig K, Cockburn J, Herlihy L, Brown C, Stahl SS, South M, McPartland JC, Kaiser MD, Schultz RT. The perception and identification of facial emotions in individuals with autism spectrum disorders using the Let's Face It! Emotion Skills Battery. J Child Psychol Psychiatry. 2012 Dec;53(12):1259-67. doi: 10.1111/j.1469-7610.2012.02571.x. Epub 2012 Jul 11. PMID 22780332
- [Background] Charlop-Christy MH, Le L, Freeman KA. A comparison of video modeling with in vivo modeling for teaching children with autism. J Autism Dev Disord. 2000 Dec;30(6):537-52. doi: 10.1023/a:1005635326276. PMID 11261466
- [Background] Gena A, Couloura S, Kymissis E. Modifying the affective behavior of preschoolers with autism using in-vivo or video modeling and reinforcement contingencies. J Autism Dev Disord. 2005 Oct;35(5):545-56. doi: 10.1007/s10803-005-0014-9. PMID 16163569
- [Background] Wilson KP. Teaching social-communication skills to preschoolers with autism: efficacy of video versus in vivo modeling in the classroom. J Autism Dev Disord. 2013 Aug;43(8):1819-31. doi: 10.1007/s10803-012-1731-5. PMID 23224593
- [Background] Klin A, Jones W, Schultz R, Volkmar F, Cohen D. Defining and quantifying the social phenotype in autism. Am J Psychiatry. 2002 Jun;159(6):895-908. doi: 10.1176/appi.ajp.159.6.895. PMID 12042174
- [Background] Landa RJ, Holman KC, O'Neill AH, Stuart EA. Intervention targeting development of socially synchronous engagement in toddlers with autism spectrum disorder: a randomized controlled trial. J Child Psychol Psychiatry. 2011 Jan;52(1):13-21. doi: 10.1111/j.1469-7610.2010.02288.x. Epub 2010 Dec 3. PMID 21126245
- [Background] Constantino, J. N., & Gruber, C. P. (2012). The Social Responsiveness Scale, Second Edition. Los Angeles, CA: Western Psychological Services.
- [Background] Lord, C., Rutter, M., DiLavore, P. C., & Risi, S. (1999). Autism Diagnostic Observation Schedule - WPS (ADOS-WPS), Los Angeles, CA: Western Psychological Services.
- [Background] Elliott C. Differential Ability Scales: Second Edition (DAS-II). San Antonio, TX: Psychological Corporation. 2007.
- [Background] Sparrow, S. S., Balla, D., Cicchetti, D. (1984). Vineland Adaptive Behavior Scales. Circle Pines, MN, American Guidance Service.
- [Background] La Greca AM, Lopez N. Social anxiety among adolescents: linkages with peer relations and friendships. J Abnorm Child Psychol. 1998 Apr;26(2):83-94. doi: 10.1023/a:1022684520514. PMID 9634131